CLINICAL TRIAL: NCT06499441
Title: Comparative Effects of Myofascial Induction Therapy Versus Gastrocnemius Pressure Release Treatment on Trigger Point Pressure Pain Threshold of the Biceps Femoris, Flexor Digitorum Brevis and Great Extensor Digitorum Muscles and Ankle ROM: Crossover Trial Study.
Brief Title: Comparative Effects of Myofascial Induction Therapy Versus Gastrocnemius Pressure Release Treatment on Trigger Point Pressure Pain Threshold in Proximal Muscles and Ankle Range of Motion.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayuben Private Clinic (Other)
Responsible Party: Principal Investigator, EVA MARIA MARTÍNEZ JIMENEZ, Physiotherapist responsible area, Mayuben Private Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2911202021420C
Record Dates: First submitted 2024-07-07; First posted 2024-07-12 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Pain Threshold; Myofascial Trigger Point; Manual Therapy; Range of Motion
Keywords: Fascia; myofascial trigger point; lower limb

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial induction in the gastrocnemius muscle (Experimental): A 3-pass shallow leg gliding technique was applied first, followed by 5 minutes of the deep myofascial calf induction technique described by Pilat.
  Interventions: Other: Myofascial induction in gastrocnemius
- Preassure release in gastrocnemius muscle (Active Comparator): Also called ischaemic pressure. Three cycles of pressure are applied to the trigger point of the gastrocnemius muscle until the pain disappears on pressure.
  Interventions: Other: Preassure release

INTERVENTIONS:
Other: Myofascial induction in gastrocnemius — A 3-pass shallow leg gliding technique was applied first, followed by 5 minutes of the deep myofascial calf induction technique described by Pilat.
  Arms: Myofascial induction in the gastrocnemius muscle
Other: Preassure release — Also called ischaemic pressure. Three cycles of pressure are applied to the trigger point of the gastrocnemius muscle until the pain disappears on pressure.
  Arms: Preassure release in gastrocnemius muscle

SUMMARY:
The aim of the study is to test the effect of myofascial induction and pre-pressure release of the grastrocnemius muscle on the proximal musculature: biceps femoris, flexor digitorum brevis and extensor digitorum grandus on the pain pre-pressure threshold variable and range of motion of ankle with knee bend and flexed

ELIGIBILITY:
Inclusion Criteria:

* Subjects from 18 to 39 years old.
* Healthy subjects with trigger point 1 of the gastrocnemius muscle in both lower limbs

Exclusion Criteria:

* Diagnosis of lower limb injury, including any tendinopathy, bursitis, ligamentous involvement, and/or fasciitis
* History of lower limb surgery or history of lower-extremity injury with residual symptoms (pain or feeling of sensations) within the last year.
* Participants could not have undergone ankle stretching or any other treatment.
* Diabetes due to possible alteration of arterial distal circulation.
* Foot deformity, cavus, and flat feet.
* Foot deformities, such as hammer toes and hallux valgus,
* Plantar corns and calluses.
* Lower limb dysfunction or chronic injury.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-08-03 (Actual)

PRIMARY OUTCOMES:
1.Threshold of pain on pressure on biceps femoris before. | Immediately before the intervention.
  The pressure at which the patient starts to feel pain with pressure is measured 3 times with an algometer. It is measured in newtons
2.Pain threshold to pressure in the extensor digitorum longus muscle before. | Immediately before the intervention.
  The pressure at which the patient starts to feel pain with pressure is measured 3 times with an algometer. It is measured in newtons
3.Pain threshold to pressure on flexor digitorum brevis muscle before. | Immediately before the intervention.
  The pressure at which the patient starts to feel pain with pressure is measured 3 times with an algometer. It is measured in newtons
4.Pain threshold on biceps femoris pressure after. | Immediately before the intervention.
  The pressure at which the patient starts to feel pain with pressure is measured 3 times with an algometer. It is measured in newtons
5.Pain threshold to pressure in the extensor digitorum longus muscle after. | Immediately before the intervention.
  The pressure at which the patient starts to feel pain with pressure is measured 3 times with an algometer. It is measured in newtons
6.Pain threshold on pressure in the flexor digitorum brevis muscle tras. | Immediately before the intervention.
  The pressure at which the patient starts to feel pain with pressure is measured 3 times with an algometer. It is measured in newtons
7. Ankle range of motion with knee extended before intervention | Immediately before the intervention.
  The joint amplitude is measured in dorsiflexion of the ankle joint with the knee extended under load and is measured with an inclinometer in degrees.
  measured in degrees.
8. Ankle range of motion with knee flexed before intervention | Immediately before the intervention.
  The joint amplitude is measured in dorsiflexion of the ankle joint with the knee flexed under load and is measured with an inclinometer in degrees.
  measured in degrees.
9. Ankle range of motion with knee extended after intervention | Immediately after the intervention.
  The joint amplitude is measured in dorsiflexion of the ankle joint with the knee extended under load and is measured with an inclinometer in degrees.
  measured in degrees.
10. Ankle range of motion with knee flexed after intervention | Immediately after the intervention.
  The joint amplitude is measured in dorsiflexion of the ankle joint with the knee flexed under load and is measured with an inclinometer in degrees.
  measured in degrees.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayuben Clinic, San Sebastián de los Reyes, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No